CLINICAL TRIAL: NCT06904573
Title: A Multicenter, Randomized Controlled Phase II Study of Evaluating the Efficacy and Safety of Immunotherapy Combined With Oral Probiotics Compound (Biolosion) in Patients With Advanced Urothelial Carcinoma
Brief Title: Probiotics in Advanced Urothelial Carcinoma
Acronym: IMPROVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Yanxia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-297
Record Dates: First submitted 2025-03-15; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Advanced Urothelial Carcinoma; Probiotics; Immunotherapy
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Gemcitabine; disitamab vedotin; enfortumab vedotin; pembrolizumab; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): Subjects in this arm will receive an oral probiotics compound (Biolosion) plus the Investigator's choice of immune checkpoint inhibitor-based (ICIs-based) therapies:
  Regimens that combine with chemotherapy agents can include but are not limited to Nab-paclitaxel, Cisplatin, Gemcitabine, Disitamab vedotin, Enfortumab Vedotin; Immune checkpoint inhibitors include but are not limited to Pembrolizumab and toripalimab.
  Interventions: Drug: Probiotics Compound (Biolosion); Drug: Nab-paclitaxel; Drug: Cisplatin; Drug: Gemcitabine; Drug: Disitamab vedotin; Drug: Enfortumab Vedotin; Drug: Pembrolizumab; Drug: Toripalimab
- Control group (Active Comparator): Subjects in this arm will receive Investigator's choice of immune checkpoint inhibitors-based (ICIs-based) therapies
  Interventions: Drug: Nab-paclitaxel; Drug: Cisplatin; Drug: Gemcitabine; Drug: Disitamab vedotin; Drug: Enfortumab Vedotin; Drug: Pembrolizumab; Drug: Toripalimab

INTERVENTIONS:
Drug: Probiotics Compound (Biolosion) — 15g, PO, qd
  Arms: Experiment group
Drug: Nab-paclitaxel — 230mg/m2, IV, days 1, 8, q3w
Drug: Cisplatin — 70mg/m2, IV, days 1-3, q3w
Drug: Gemcitabine — 1.2g/m2, IV, days 1, 8, q3w
Drug: Disitamab vedotin — 2.5mg/kg, IV, q2w
Drug: Enfortumab Vedotin — 1.25mg/kg, IV, days 1, 8, q3w
Drug: Pembrolizumab — 200mg, IV, q3w
Drug: Toripalimab — 240mg, IV, q3w

SUMMARY:
This is a multicenter, randomized, controlled phase II Study of evaluating the efficacy and safety of immunotherapy combined with probiotics compound (Biolosion) in patients with advanced urothelial carcinoma.

DETAILED DESCRIPTION:
This multicenter, randomized phase II trial is designed to study the efficacy and safety of probiotics compound (Biolosion) Immunotherapy of the physician's choice (IPC) plus versus IPC in patients with advanced urothelial carcinoma (aUC). Pervious received platinum-based therapies, previous received Immune checkpoint inhibitors, and the treatment lines will stratify randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study must meet all of the following criteria:

  1. Aged 18 or above;
  2. Histologically or cytologically confirmed locally advanced inoperable (such as T4b, or N2-3) or metastatic urothelial carcinoma, including bladder, ureter, renal pelvis and urethra;
  3. Patients who have received previous treatment with immune checkpoint inhibitors (PD-1/PD-L1 monoclonal antibodies) are allowed;
  4. According to RECIST1.1 standard, there is at least one measurable target lesion;
  5. ECOG score ≤2;
  6. Good bone marrow, kidney (serum creatinine clearance calculated by CG formula> 30 mL/min), liver and coagulation function:
  7. Expected survival period ≥ 6 months;
  8. The patient understands the research procedures and signs the informed consent form in writing to indicate his/her agreement to participate in the study;
  9. Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 7 days before the first dose of study drug (Cycle 1, Day 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required.
  10. If there is a risk of pregnancy, male and female patients should use highly effective contraception (i.e., a method with a failure rate of less than 1% per year) and continue for at least 180 days after stopping the trial treatment.

Exclusion Criteria:

* Any of the following will be considered as meeting the exclusion criteria of the study:

  1. Patients with locally advanced disease may receive local radical treatment;
  2. History of clinically symptomatic cardiovascular, liver, respiratory, renal, hematoendocrine, or neuropsychiatric diseases;
  3. Clear brain/meningeal metastasis;
  4. Peripheral neuropathy >1 degree;
  5. Patients who have received anti-tumor monoclonal antibody treatment within 4 weeks before the start of the study, or have received other anti-tumor drug treatment and have not recovered from adverse events/reactions;
  6. Participated in any investigational drug treatment within 4 weeks before the start of treatment;
  7. Patients who had received axial bone radiotherapy within 4 weeks before the start of the study or had not recovered from adverse reactions caused by previous radiotherapy;
  8. Known severe allergic reaction to the study drug, its active ingredients and/or any excipients;
  9. Patients diagnosed with immunodeficiency or receiving systemic glucocorticoids or any other form of immunosuppressive therapy within 7 days before the first dose of the study; physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent drugs) are allowed;
  10. Active autoimmune diseases requiring systemic treatment (such as the use of disease-modifying drugs, corticosteroids, or immunosuppressants) occurred within 2 years before the first dose. Replacement therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatment; a history of non-infectious pneumonia requiring glucocorticoid treatment within 1 year before the first dose or current interstitial lung disease;
  11. Received solid organ or blood system transplantation;
  12. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive). Untreated active hepatitis B;
  13. Untreated active hepatitis B; Note: Hepatitis B subjects who meet the following criteria are also eligible for inclusion: HBV viral load must be <1000 copies/ml (200 IU/ml) before the first dose, and subjects should receive anti-HBV treatment during the entire study chemotherapy treatment to avoid viral reactivation. For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), preventive anti-HBV treatment is not required, but viral reactivation needs to be closely monitored;
  14. Subjects with active HCV infection (HCV antibody positive and HCV-RNA level above the detection limit) received live vaccine within 30 days before the first dose (Cycle 1, Day 1);
  15. A history of other malignant tumors in the past 5 years, excluding cured non-malignant melanoma of the skin, cervical carcinoma in situ, and incidentally discovered prostate cancer (stage lower than T2N0M0, Gleason score <7, or undetectable PSA);
  16. Medical history or disease evidence, abnormal treatment or laboratory test values, or other conditions that the researcher considers unsuitable for enrollment that may interfere with the trial results or prevent the subject from fully participating in the study;
  17. Breastfeeding women
  18. People with chronic diseases who need to take antibiotics for a long time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Within approximately 48 months
  Progression-Free Survival (PFS) is defined as the time from randomization to the first documented disease progression, as determined by RECIST v1.1, or death from any cause, whichever occurs first. Disease progression will be assessed by independent radiologic review. Patients without documented progression or death at the time of analysis will be censored at their last tumor assessment date.

SECONDARY OUTCOMES:
Overall Survival (OS) | Within approximately 48 months
  Overall Survival (OS) is defined as the time from randomization to death from any cause. Participants still alive at the time of analysis will be censored at the date of the last follow-up.
Objective Response Rate (ORR) | Within approximately 48 months
  Objective Response Rate (ORR) is defined as the proportion of participants achieving a complete response (CR) or partial response (PR) as determined by RECIST v1.1 criteria, based on radiologic assessment. Responses will be confirmed by at least one subsequent imaging assessment.
Disease Control Rate (DCR) | Within approximately 48 months
  Disease Control Rate (DCR) is defined as the proportion of participants achieving a complete response (CR), partial response (PR), or stable disease (SD) for at least 6 weeks after treatment initiation, based on RECIST v1.1 criteria.
Time to Response (TTR) | Within approximately 48 months
  Time to Response (TTR) is defined as the time from randomization to the first occurrence of a confirmed objective response (CR or PR) as determined by RECIST v1.1 criteria.
Duration of Response (DOR) | Within approximately 48 months
  Duration of Response (DOR) is defined as the time from the first documented objective response (CR or PR) to disease progression or death, whichever occurs first, based on RECIST v1.1 criteria.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Within approximately 48 months
  The number of participants who experience treatment-related adverse events (AEs) will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. AEs will be graded on a scale from Grade 1 (mild) to Grade 5 (death related to AE). The severity, frequency, and type of AEs will be recorded and summarized. The results will be presented as the total number and percentage of participants experiencing any treatment-related AE, as well as a breakdown by AE grade and type. Treatment-related AEs will be determined by the investigator's clinical judgment based on available data.

OTHER OUTCOMES:
Analysis of the microbiota | Baseline, through study completion, an average of 48 months
  The stool samples of participants before and after treatment were collected and analyzed by 16S rRNA and were used to investigate the changes in the diversity of microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Shi, Doctor, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Sun yat-sen university cancer center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical and privacy concerns.

REFERENCES:
- [Background] Dizman N, Meza L, Bergerot P, Alcantara M, Dorff T, Lyou Y, Frankel P, Cui Y, Mira V, Llamas M, Hsu J, Zengin Z, Salgia N, Salgia S, Malhotra J, Chawla N, Chehrazi-Raffle A, Muddasani R, Gillece J, Reining L, Trent J, Takahashi M, Oka K, Higashi S, Kortylewski M, Highlander SK, Pal SK. Nivolumab plus ipilimumab with or without live bacterial supplementation in metastatic renal cell carcinoma: a randomized phase 1 trial. Nat Med. 2022 Apr;28(4):704-712. doi: 10.1038/s41591-022-01694-6. Epub 2022 Feb 28. PMID 35228755
- [Background] Miyake M, Oda Y, Owari T, Iida K, Ohnishi S, Fujii T, Nishimura N, Miyamoto T, Shimizu T, Ohnishi K, Hori S, Morizawa Y, Gotoh D, Nakai Y, Torimoto K, Tanaka N, Fujimoto K. Probiotics enhances anti-tumor immune response induced by gemcitabine plus cisplatin chemotherapy for urothelial cancer. Cancer Sci. 2023 Mar;114(3):1118-1130. doi: 10.1111/cas.15666. Epub 2022 Nov 30. PMID 36398663
- [Background] Messaoudene M, Pidgeon R, Richard C, Ponce M, Diop K, Benlaifaoui M, Nolin-Lapalme A, Cauchois F, Malo J, Belkaid W, Isnard S, Fradet Y, Dridi L, Velin D, Oster P, Raoult D, Ghiringhelli F, Boidot R, Chevrier S, Kysela DT, Brun YV, Falcone EL, Pilon G, Onate FP, Gitton-Quent O, Le Chatelier E, Durand S, Kroemer G, Elkrief A, Marette A, Castagner B, Routy B. A Natural Polyphenol Exerts Antitumor Activity and Circumvents Anti-PD-1 Resistance through Effects on the Gut Microbiota. Cancer Discov. 2022 Apr 1;12(4):1070-1087. doi: 10.1158/2159-8290.CD-21-0808. PMID 35031549
- [Background] Sivan A, Corrales L, Hubert N, Williams JB, Aquino-Michaels K, Earley ZM, Benyamin FW, Lei YM, Jabri B, Alegre ML, Chang EB, Gajewski TF. Commensal Bifidobacterium promotes antitumor immunity and facilitates anti-PD-L1 efficacy. Science. 2015 Nov 27;350(6264):1084-9. doi: 10.1126/science.aac4255. Epub 2015 Nov 5. PMID 26541606
- [Background] Li WT, Iyangar AS, Reddy R, Chakladar J, Bhargava V, Sakamoto K, Ongkeko WM, Rajasekaran M. The Bladder Microbiome Is Associated with Epithelial-Mesenchymal Transition in Muscle Invasive Urothelial Bladder Carcinoma. Cancers (Basel). 2021 Jul 21;13(15):3649. doi: 10.3390/cancers13153649. PMID 34359550
- [Background] Grande E, G.M., Arranz Arija JA, et al., IMvigor130: a phase III study of atezolizumab with or without platinum-based chemotherapy in previously untreated metastatic urothelial carcinoma. Presented at: . ESMO Congress; , 2019 Abstract LBA14.
- [Background] Lichtenegger FS, Rothe M, Schnorfeil FM, Deiser K, Krupka C, Augsberger C, Schluter M, Neitz J, Subklewe M. Targeting LAG-3 and PD-1 to Enhance T Cell Activation by Antigen-Presenting Cells. Front Immunol. 2018 Feb 27;9:385. doi: 10.3389/fimmu.2018.00385. eCollection 2018. PMID 29535740
- [Background] Champiat S, Dercle L, Ammari S, Massard C, Hollebecque A, Postel-Vinay S, Chaput N, Eggermont A, Marabelle A, Soria JC, Ferte C. Hyperprogressive Disease Is a New Pattern of Progression in Cancer Patients Treated by Anti-PD-1/PD-L1. Clin Cancer Res. 2017 Apr 15;23(8):1920-1928. doi: 10.1158/1078-0432.CCR-16-1741. Epub 2016 Nov 8. PMID 27827313
- [Background] Vaughn DJ, Bellmunt J, Fradet Y, Lee JL, Fong L, Vogelzang NJ, Climent MA, Petrylak DP, Choueiri TK, Necchi A, Gerritsen W, Gurney H, Quinn DI, Culine S, Sternberg CN, Mai Y, Li H, Perini RF, Bajorin DF, de Wit R. Health-Related Quality-of-Life Analysis From KEYNOTE-045: A Phase III Study of Pembrolizumab Versus Chemotherapy for Previously Treated Advanced Urothelial Cancer. J Clin Oncol. 2018 Jun 1;36(16):1579-1587. doi: 10.1200/JCO.2017.76.9562. Epub 2018 Mar 28. PMID 29590008
- [Background] Powles T, O'Donnell PH, Massard C, Arkenau HT, Friedlander TW, Hoimes CJ, Lee JL, Ong M, Sridhar SS, Vogelzang NJ, Fishman MN, Zhang J, Srinivas S, Parikh J, Antal J, Jin X, Gupta AK, Ben Y, Hahn NM. Efficacy and Safety of Durvalumab in Locally Advanced or Metastatic Urothelial Carcinoma: Updated Results From a Phase 1/2 Open-label Study. JAMA Oncol. 2017 Sep 14;3(9):e172411. doi: 10.1001/jamaoncol.2017.2411. Epub 2017 Sep 14. PMID 28817753
- [Background] Sharma P, Retz M, Siefker-Radtke A, Baron A, Necchi A, Bedke J, Plimack ER, Vaena D, Grimm MO, Bracarda S, Arranz JA, Pal S, Ohyama C, Saci A, Qu X, Lambert A, Krishnan S, Azrilevich A, Galsky MD. Nivolumab in metastatic urothelial carcinoma after platinum therapy (CheckMate 275): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2017 Mar;18(3):312-322. doi: 10.1016/S1470-2045(17)30065-7. Epub 2017 Jan 26. PMID 28131785
- [Background] Petrylak DP, Powles T, Bellmunt J, Braiteh F, Loriot Y, Morales-Barrera R, Burris HA, Kim JW, Ding B, Kaiser C, Fasso M, O'Hear C, Vogelzang NJ. Atezolizumab (MPDL3280A) Monotherapy for Patients With Metastatic Urothelial Cancer: Long-term Outcomes From a Phase 1 Study. JAMA Oncol. 2018 Apr 1;4(4):537-544. doi: 10.1001/jamaoncol.2017.5440. PMID 29423515
- [Background] Sio TT, Ko J, Gudena VK, Verma N, Chaudhary UB. Chemotherapeutic and targeted biological agents for metastatic bladder cancer: a comprehensive review. Int J Urol. 2014 Jul;21(7):630-7. doi: 10.1111/iju.12407. Epub 2014 Jan 23. PMID 24455982
- [Background] Lin CC, Hsu CH, Huang CY, Keng HY, Tsai YC, Huang KH, Cheng AL, Pu YS. Gemcitabine and ifosfamide as a second-line treatment for cisplatin-refractory metastatic urothelial carcinoma: a phase II study. Anticancer Drugs. 2007 Apr;18(4):487-91. doi: 10.1097/CAD.0b013e3280126603. PMID 17351402
- [Background] Sweeney CJ, Roth BJ, Kabbinavar FF, Vaughn DJ, Arning M, Curiel RE, Obasaju CK, Wang Y, Nicol SJ, Kaufman DS. Phase II study of pemetrexed for second-line treatment of transitional cell cancer of the urothelium. J Clin Oncol. 2006 Jul 20;24(21):3451-7. doi: 10.1200/JCO.2005.03.6699. PMID 16849761
- [Background] Vaughn DJ, Broome CM, Hussain M, Gutheil JC, Markowitz AB. Phase II trial of weekly paclitaxel in patients with previously treated advanced urothelial cancer. J Clin Oncol. 2002 Feb 15;20(4):937-40. doi: 10.1200/JCO.2002.20.4.937. PMID 11844814
- [Background] Bellmunt J, Theodore C, Demkov T, Komyakov B, Sengelov L, Daugaard G, Caty A, Carles J, Jagiello-Gruszfeld A, Karyakin O, Delgado FM, Hurteloup P, Winquist E, Morsli N, Salhi Y, Culine S, von der Maase H. Phase III trial of vinflunine plus best supportive care compared with best supportive care alone after a platinum-containing regimen in patients with advanced transitional cell carcinoma of the urothelial tract. J Clin Oncol. 2009 Sep 20;27(27):4454-61. doi: 10.1200/JCO.2008.20.5534. Epub 2009 Aug 17. PMID 19687335
- [Background] De Santis M, Bellmunt J, Mead G, Kerst JM, Leahy M, Maroto P, Gil T, Marreaud S, Daugaard G, Skoneczna I, Collette S, Lorent J, de Wit R, Sylvester R. Randomized phase II/III trial assessing gemcitabine/carboplatin and methotrexate/carboplatin/vinblastine in patients with advanced urothelial cancer who are unfit for cisplatin-based chemotherapy: EORTC study 30986. J Clin Oncol. 2012 Jan 10;30(2):191-9. doi: 10.1200/JCO.2011.37.3571. Epub 2011 Dec 12. PMID 22162575
- [Background] von der Maase H, Hansen SW, Roberts JT, Dogliotti L, Oliver T, Moore MJ, Bodrogi I, Albers P, Knuth A, Lippert CM, Kerbrat P, Sanchez Rovira P, Wersall P, Cleall SP, Roychowdhury DF, Tomlin I, Visseren-Grul CM, Conte PF. Gemcitabine and cisplatin versus methotrexate, vinblastine, doxorubicin, and cisplatin in advanced or metastatic bladder cancer: results of a large, randomized, multinational, multicenter, phase III study. J Clin Oncol. 2000 Sep;18(17):3068-77. doi: 10.1200/JCO.2000.18.17.3068. PMID 11001674
- [Background] Abida W, Bajorin DF, Rosenberg JE. First-line treatment and prognostic factors of metastatic bladder cancer for platinum-eligible patients. Hematol Oncol Clin North Am. 2015 Apr;29(2):319-28, ix-x. doi: 10.1016/j.hoc.2014.10.005. Epub 2014 Dec 15. PMID 25836937
- [Background] Chen W, Zheng R, Zeng H, Zhang S, He J. Annual report on status of cancer in China, 2011. Chin J Cancer Res. 2015 Feb;27(1):2-12. doi: 10.3978/j.issn.1000-9604.2015.01.06. PMID 25717220